CLINICAL TRIAL: NCT04647734
Title: The Protective Potential of Exercise Training on the Cardiopulmonary Morbidity After COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Regitse Christensen, Principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H-20033733 v.2
Record Dates: First submitted 2020-11-25; First posted 2020-12-01 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: COVID-19, SARS-CoV2
MeSH Terms: conditions — COVID-19 | interventions — High-Intensity Interval Training; Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity interval training (Experimental): The experimental group will on top of standard care undergo a 12 weeks supervised exercise high intensity interval exercise training on an ergometer bike three times a week for 38 minutes. The specific intervals will be determined from our ongoing pilot study (NCT04549337)
  Interventions: Behavioral: High intensity interval training
- Control group (Active Comparator): This group will be allocated to standard care and therefore no supervised exercise regimen.
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: High intensity interval training — 12 weeks of high intensity interval training on exercise bike for 38 minutes 3 times a week
  Arms: High intensity interval training
Behavioral: Standard care — standard care after discharge from hospital (control group)
  Arms: Control group

SUMMARY:
40 COVID-19 survivors that have been discharged from the hospital will be included in this investigator-blinded randomised study with a 12-week exercise intervention. Patients will be 1:1 block-randomised by sex to either a supervised high intensity interval-based exercise group or standard care (control group).

DETAILED DESCRIPTION:
40 patients will be recruited and undergo baseline testing, including examination, biochemistry, ECG, DXA, OGTT, Pulmonary function, VO2max, RM, plasma volume, AX3, CGM, echocardiography, cardiac MRI.

After baseline testing, participants will be randomly allocated into one group receiving standard of care (control group) or a group performing supervised high-intensity interval training three times a week over a period of 12 weeks. The randomization procedure involves a computer-generated block randomization schedule in a ratio of 1:1 stratified by sex by an independent person. Following the 12-week intervention period, both groups will complete a series of follow-up tests (as baseline testing). A 1-year follow-up experimental day is also planned in order to evaluate fitness, cardiac and pulmonary structure and function.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years
* A laboratory-confirmed initial positive test followed by one negative tests of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) ≤ 6 months after hospital discharge
* ≤10 L oxygen requirement during hospitalization

Exclusion Criteria:

* Present atrial fibrillation
* Diagnosed with acute myocarditis
* Health conditions that prevent participating in the exercise intervention
* Patients who cannot undergo MR scans (e.g. kidney disease or metallic implants)
* Treatment with IL-6 receptor antagonists (tocilizumab, kevzara) within the last month due to drug interference with the cardiopulmonary exercise adaptations.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular mass | Through study completion, an average of 12 months
  measured by MRI scan
Change in right ventricular volume | Through study completion, an average of 12 months
  measured by MRI scan

SECONDARY OUTCOMES:
Stroke volume | Through study completion, an average of 12 months
  Structural cardiac parameter: measured by MRI scan and echocardiography
end-diastolic volume | Through study completion, an average of 12 months
  Structural cardiac parameter: measured by MRI scan and echocardiography
IVS thickness (intact ventricular septum) | Through study completion, an average of 12 months
  Structural cardiac parameter: measured by MRI scan and echocardiography
LVID (left ventricular internal dimensions) | Through study completion, an average of 12 months
  Structural cardiac parameter: measured by MRI scan and echocardiography
PWT (posterior wall thickness) | Through study completion, an average of 12 months
  Structural cardiac parameter: measured by MRI scan and echocardiography
LAVI (left atrial volume index) | Through study completion, an average of 12 months
  Structural cardiac parameter: measured by MRI scan and echocardiography
LVEF | Through study completion, an average of 12 months
  Functional cardiac parameters: measured by MRI scan and echocardiography
Global longitudinal strain | Through study completion, an average of 12 months
  Functional cardiac parameters: measured by MRI scan and echocardiography
E/A ratio | Through study completion, an average of 12 months
  Functional cardiac parameters: measured by MRI scan and echocardiography
E´ | Through study completion, an average of 12 months
  Functional cardiac parameters: measured by MRI scan and echocardiography
RV volumes | Through study completion, an average of 12 months
  Functional cardiac parameters: measured by MRI scan and echocardiography
RVEF | Through study completion, an average of 12 months
  Functional cardiac parameters: measured by MRI scan and echocardiography
TAPSE | Through study completion, an average of 12 months
  Functional cardiac parameters: measured by MRI scan and echocardiography
Change in maximal tricuspid regurgitation velocity and pressure gradient | Through study completion, an average of 12 months
  Functional cardiac parameters: measured by MRI scan and echocardiography
RV s´ | Through study completion, an average of 12 months
  Functional cardiac parameters: measured by MRI scan and echocardiography
Peak E velocity | Through study completion, an average of 12 months
  Functional cardiac parameters: measured by MRI scan and echocardiography
Peak A velocity | Through study completion, an average of 12 months
  Functional cardiac parameters: measured by MRI scan and echocardiography
Septal e´ | Through study completion, an average of 12 months
  Functional cardiac parameters: measured by MRI scan and echocardiography
Lateral e´ | Through study completion, an average of 12 months
  Functional cardiac parameters: measured by MRI scan and echocardiography
E/e´ septal | Through study completion, an average of 12 months
  Functional cardiac parameters: measured by MRI scan and echocardiography
E/e´ lateral | Through study completion, an average of 12 months
  Functional cardiac parameters: measured by MRI scan and echocardiography
Cardiac inflammation | Through study completion, an average of 12 months
  measured with gadolinium and MRI scan
Vascular dysfunction | Through study completion, an average of 12 months
  measured with gadolinium and MRI scan
Extracellular volume | Through study completion, an average of 12 months
  measured with gadolinium and MRI scan
Diffuse fibrotic changes | Through study completion, an average of 12 months
  measured with gadolinium and MRI scan
Blood and plasma volume | Through study completion, an average of 12 months
  changes
Body composition analysis measured with DXA | Through study completion, an average of 12 months
  easuring Lean mass, Fat mass and BMD
Cardiorespiratory fitness | Through study completion, an average of 12 months
  Measured with an incremental VO2 protocol on exercise bike
Dynamic spirometri | Through study completion, an average of 12 months
  Pulmonary function testing
Whole body plethymography | Through study completion, an average of 12 months
  Pulmonary function testing
Diffusion capacity | Through study completion, an average of 12 months
  Pulmonary function testing
Oral glucose tolerance test | 2 hours at baseline and same after intervention
  75g of glucose taken while fasting
Continuous glucose monitoring | 3 days at baseline and same after intervention
  Three days of continuous glucose monitoring (CGM) is performed using enzyme-coated electrodes (iPro MMT- 7745WW; Medtronic, Northridge, CA, USA) placed subcutaneously in the abdominal wall. For calibration of the CGM system, finger-prick blood glucose measurements are performed by the participant four times daily.
Axial accelerometer-based physical activity monitors | 4 days at baseline and same after intervention
  Free-living physical activity is measured using axial accelerometer-based physical activity monitors (AX3; Axivity, Newcastle upon Tyne, UK) for a 4-day period
Blood samples analysed for markers related to low grade inflammation | Through study completion, an average of 12 months
  Including high-sensitivity C-reactive protein, tumour necrosis factor-α, IL-1RA, interferon-γ and interleukins (IL-6, IL-10 and others)
  Following an overnight fast (10 hours), blood samples, are collected and processed by a trained laboratory technician and analysed according to standard procedures. Plasma is stored at - 80 °C prior to analysis.
Blood samples analysed for markers related to cardiometabolic biomarkers. | Through study completion, an average of 12 months
  Including total troponins, D-dimer, creatinine kinase, total cholesterol, high-density lipoprotein, low-density lipoprotein, triglycerides, glycated haemoglobin, fasting insulin, fasting plasma glucose, pro-brain natriuretic peptide, haematology, electrolytes and liver and renal status.
  Following an overnight fast (10 hours), blood samples, are collected and processed by a trained laboratory technician and analysed according to standard procedures. Plasma is stored at - 80 °C prior to analysis.
SF-36, King´s Brief Interstitial Lung Disease Questionnaire, Post-COVID-19 Functional Status | Through study completion, an average of 12 months
  Questionnaires on quality of life will be filled in on baseline and after the intervention
King´s Brief Interstitial Lung Disease Questionnaire | Through study completion, an average of 12 months
  Questionnaires on quality of life will be filled in on baseline and after the intervention
Post-COVID-19 Functional Status | Through study completion, an average of 12 months
  Questionnaires on quality of life will be filled in on baseline and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Regitse Christensen, MD, PhD, Principal Investigator — Center for Physical Activity Research, Rigshospitalet
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Rasmussen IE, Foged F, Bjorn Budde J, Rasmussen RS, Rasmussen V, Lyngbaek M, Jonck S, Krogh-Madsen R, Lindegaard B, Ried-Larsen M, Jorgensen PG, Lund MAV, Kober L, Vejlstrup N, Pedersen BK, Berg RMG, Christensen RH. Protective potential of high-intensity interval training on cardiac structure and function after COVID-19: protocol and statistical analysis plan for an investigator-blinded randomised controlled trial. BMJ Open. 2021 Nov 18;11(11):e048281. doi: 10.1136/bmjopen-2020-048281. PMID 34794987